CLINICAL TRIAL: NCT00456326
Title: A 3 Year Retrospective Heparin Induced Thrombocytopenia Registry (HIT) at Brigham and Women's Hospital.
Brief Title: Heparin-Induced Thrombocytopenia Registry
Acronym: HIT
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Samuel Z. Goldhaber, MD, Brigham and Women's Hospital
Other Study IDs: 2005-P-001941
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Heparin-Induced Thrombocytopenia
Keywords: Heparin; Unfractionated Heparin; Low Molecular Weight Heparin; Anticoagulation; Thrombocytopenia; Thrombosis; Venous Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Thrombocytopenia; Thrombosis; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIT Patients: Patients at Brigham and Women's Hospital diagnosed with Heparin Induced Thrombocytopenia.

SUMMARY:
The purpose of the Heparin Induced Thrombocytopenia Registry is to explore the frequency of heparin-induced thrombocytopenia (HIT) at Brigham and Women's Hospital and to assess its mortality rate. Retrospective 3 years, looking forward prospectively.

DETAILED DESCRIPTION:
Heparin-induced thrombocytopenia (HIT) is an immune-mediated adverse drug reaction with potentially fatal complications of venous and arterial thrombosis.

HIT with thrombosis causes prolonged hospital length of stay and is associated with catastrophic outcomes such as extremity amputation as well as death. The fear of HIT has led to some proposals to minimize hospital use of unfractionated heparin (UFH) and low molecular weight heparin (LMWH) and to substitute other anticoagulants that have not been reported to cause HIT. Therefore, the frequency of confirmed HIT and the frequency of determining whether UFH or LMWH is the causative agent urgently require further investigation.

At BWH, we have placed patient safety at a premium. We have a Patient Safety Committee and a Patient Safety Officer. HIT has been identified as one of the primary problems requiring urgent policy decisions. Consequently, we have formed a multi-disciplinary team of physicians, pharmacists, nurses and physician's assistants to improve safe medication practices for patients receiving anticoagulation.

Our primary objectives are to establish an HIT registry which will provide information on:

1. Incidence of HIT associated with UFH and LMWH
2. Outcomes of patients with HIT
3. Adverse events associated with alternative anticoagulants used to treat HIT

We will obtain data with respect to: Drug, Dose, Route of administration, Duration of therapy, Platelet count, Platelet nadir, Co-morbidities (Coronary Artery Disease, Diabetes Mellitus, Myocardial Infarction, Hypertension, Pulmonary Disease, Chronic Renal Failure, Malignancy, Liver Disease, Surgery, Sepsis), Baseline characteristics (Age, Sex, Weight), Pregnancy status, Serum Creatinine, AST, ALT, Hematocrit, Hemoglobin, Venous and Arterial Thrombotic events (DVT, PE, CVC), 30-day mortality rate, alternative anticoagulant therapy, and duration of therapy.

Time and Method of Data Collection:

Chart Review for the duration of hospitalization: Hemorrhagic event, Thrombotic events, and 30-day Mortality Rate.

ELIGIBILITY:
All patients hospitalized at BWH who have a PF4-Positive antibody test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Heparin Induced Thrombocytopenia
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2005-10; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Incidence of HIT associated with UFH and LMWH | 30 Days
Outcomes of patients with HIT | 30 Days
Adverse events associated with alternative anticoagulants used to treat HIT | 30 Days

SECONDARY OUTCOMES:
Mortality | 30 Days
Hemorrhagic Events | 30 Days
Thrombotic Events | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Z. Goldhaber, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Baroletti SA, Goldhaber SZ. Heparin-induced thrombocytopenia. Circulation. 2006 Aug 22;114(8):e355-6. doi: 10.1161/CIRCULATIONAHA.106.632653. No abstract available. PMID 16923760
- See also: North American Thrombosis Forum — http://www.NATFonline.org